CLINICAL TRIAL: NCT07001605
Title: Comparing the Quality of Recovery of Erector Spinae Block Versus Ketamine-based Multimodal Analgesia Protocol in Lumber Decompressive Surgery: a Randomized Controlled Trial
Brief Title: Erector Spinae Block Vs Ketamine-based Multimodal Analgesia Protocol in Lumber Decompressive Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-18-2025
Record Dates: First submitted 2025-05-15; First posted 2025-06-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Spinal Decompression; Analgesia; Erector Spinae Plane Block; Ketamine
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ketamine group (Active Comparator): Patients will be receiving ketamine bolus then continuous infusion and local wound infiltration at the end of the surgery.
  Interventions: Drug: ketamine; Other: Wound infiltration
- ESPB group (Active Comparator): Patients will be receiving erector spinae plane block
  Interventions: Other: Erector Spinae Plane Block

INTERVENTIONS:
Drug: ketamine — after induction of anesthesia, patients will receive ketamine bolus of 0.5 mL/kg followed by continuous infusion of 0.12 mL/k/hr until the end of surgical procedure.
  Arms: ketamine group
Other: Erector Spinae Plane Block — after induction of anesthesia, patients will receive ultrasound guided ESPB. A total of 40 mL of 0.25% bupivacaine will be injected bilaterally at the level of transverse process opposing to the mid-point of the planned incision.
  Arms: ESPB group
Other: Wound infiltration — wound infiltration at the end of the surgery before the closure of fascia and subcutaneous tissues using a total of 20 ml of 0.25% bupivacaine
  Arms: ketamine group

SUMMARY:
The aim of this study is to compare the quality of recovery of the erector spinae plane block (ESPB) versus ketamine-based multimodal analgesia regimen after spine decompressive surgery.

DETAILED DESCRIPTION:
Preoperatively, standard monitors will be attached (electrocardiogram, noninvasive blood pressure, and pulse oximetry) and intravenous access will be obtained. Dexamethasone will be administered at dose of 4 mg as an antiemetic prophylaxis.

Thirty min before induction of anesthesia all patients will receive 15 mg ketorolac and 1 gm paracetamol intravenously.

General anesthesia will be induced by 1 mcg/kg fentanyl and 2 mg/kg propofol titrated till loss of verbal response. Tracheal intubation will be facilitated by 0.5 mg/kg atracurium. General anesthesia will be maintained by isoflurane (end-tidal isoflurane concentration of 1-1.2%) in air-oxygen admixture.

Fentanyl boluses of 50 mcg will be given in case of inadequate analgesia (heart rate and or systolic blood pressure increase by 20% from the baseline in absence of other causes) Intraoperative hemodynamic management will be according to the discretion of the attending anesthetist.

Postoperatively, all Patients will receive oral 1 gm of paracetamol every 6 h and 400 mg ibuprofen every 8 h.

Pain assessments using NRS (Numerical Rating Scale) at rest and during movement at 0.5 , 4, 10, 18 and 24 h postoperatively. If NRS score is > 3, intravenous nalbuphine 0.1 mg/kg (lean body weight) titrated to response will be given (maximum single dose is 20 mg and maximum daily dose is 160 mg).

Intravenous ondansetron 4 mg will be given to treat nausea or vomiting if occurs.

At the end of 24 h postoperatively, patient's quality of recovery will be assessed using QoR-15 questionnaire and patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status of I-III
* scheduled for open lumber decompression surgery for degenerative stenosis or trauma involving 1or 2 levels without fusion.

Exclusion Criteria:

* Refusal to participate
* Contraindication for peripheral regional anesthesia such as infection and coagulopathy.
* Inability to comprehend the Numeric Rating Scale (NRS) or Patients who has cognitive function impairment
* Preoperative renal or hepatic insufficiency
* History of Opioid abuse.
* Allergy to any of the study drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
quality of recovery | 24 hour to 25 hour after surgery
  using the QoR-15 questionnaire

SECONDARY OUTCOMES:
pain assessment | 30 minutes postoperatively till 24 hours postoperatively
  numerical rating scale
nalbuphine requirement | 30 minutes postoperatively till 24 hours postoperatively
  mg
time to rescue analgesia | 30 minutes postoperatively till 24 hours postoperatively
  hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data used for statistical analysis are available from the PI upon reasonable request